CLINICAL TRIAL: NCT06422936
Title: SPOTLIGHT 204: A Multicenter, Phase 2b, Open-label, Non-randomized, Clinical Trial to Evaluate Safety, Tolerability and Preliminary Efficacy of Intra-lesional BO-112 in Patients With Resectable Primary Low and High Risk Basal Cell Carcinoma
Brief Title: Clinical Trial to Evaluate BO-112 in Patients With Basal Cell Carcinoma (BCC)
Acronym: SPOTLIGHT204
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Highlight Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BOT-112-204
Record Dates: First submitted 2024-05-13; First posted 2024-05-21 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — BO-112

STUDY DESIGN:
Intervention Model Description: Parallel group design with same treatment and study procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort I (Experimental): patients with low risk nodular BCC
  Interventions: Drug: BO-112
- Cohort II (Experimental): patients with high risk BCC
  Interventions: Drug: BO-112

INTERVENTIONS:
Drug: BO-112 — Noncoding double-stranded (ds) RNA based on polyinosinic-polycytidylic acid (Poly I:C), formulated with polyethylenimine (PEI) for intra-lesional injection

SUMMARY:
This is a multicenter, phase 2b, open-label, non-randomized, clinical trial to evaluate safety, tolerability, pharmacodynamics and preliminary efficacy of intra-lesional BO-112 in patients with resectable primary low and high risk basal cell carcinoma.

* primary endpoint is visual and pathological response [at surgery] on patient level assessed by central review
* secondary endpoints are

  1. Occurrence of adverse events (AEs), serious adverse events (SAEs), and AEs leading to discontinuation or death on patient level.
  2. Pathological response [at surgery] on patient level assessed by the investigator and central review, respectively, and visual response [during the study and at surgery] on patient level assessed by the investigator and central review, respectively.
  3. Recurrence [at 12 and 24 months] after surgery on patient level assessed by the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥ 18 years old [or the legal age of consent in the jurisdiction in which the study is taking place], at the time of signing the informed consent.

   Type of Participant and Disease Condition
2. Has primary resectable low or high risk basal cell carcinoma according to the protocol definition
3. Has diagnostic punch biopsy of all lesions intended for injection available prior to the first dose of BO-112.
4. Has adequate organ function defined as defined per protocol
5. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of study drug.
6. Women of childbearing potential must be willing to use two effective methods of birth control while treated with BO-112 and for 4 weeks after the last treatment. The two forms of birth control authorized are defined as the use of a barrier method of contraception (condom with spermicide) in association with one of the following methods of birth control: bilateral tubal ligation; combined oral contraceptives (estrogens and progesterone) or implanted or injectable contraceptives from the time of informed consent.
7. Male patients with female partners of childbearing potential must be willing to use two adequate contraception methods while treated with BO-112 and for 4 weeks after treatment completion.

   Informed Consent
8. Capable of giving signed informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
9. Able and willing to comply with all study requirements, including surgical removal of lesion/lesion site at completion of study.

Exclusion Criteria:

1. Has history of hypersensitivity to BO-112 or its excipients/vehicle. 2. Has any BCC lesion(s) in site of prior radiation and/or any BCC lesion(s) within 2 cm of the open eyelid margins 4. Has Gorlin's syndrome 5. Has clinically active or uncontrolled skin disease or tattoos that would interfere with evaluation of the area surrounding the target lesion 6. Has another malignant disease requiring treatment 7. Has a history of immunological disorder, severe allergic reaction, moderate or severe asthma or known history of anaphylaxis or any other serious adverse reactions to the investigational products.

8. Female participants: lactating or pregnant. 9. Has received a live vaccine or messenger ribonucleic acid (mRNA) Corona virus disease (COVID) vaccine within 7 days prior to the first dose of study drug or has a vaccination planned during treatment with BO-112 and within 7 days after the last study drug administration.

10. Is immunocompromised. Systemic corticosteroids at >10 mg/day prednisone or equivalent within 1 week prior to the first dose of BO-112.

11. Has any prior systemic anti-lesion therapy or local treatment for study lesions prior to first dose; any chemotherapy or immunotherapy for any other malignancy within 24 months prior to the first dose of BO-112.

12. Has any experimental or investigational agents within one month of first BO-112 injection.

13. Has received or is expected to receive treatment with psoralen plus ultraviolet A (UVA) or ultraviolet B (UVB) therapy within 6 months prior to the first dose of BO-112.

14. Requires / or has used topical products within 5 cm of a treatment-targeted BCC lesion or systemic therapies that might interfere with the evaluation of the study medication during the study.

15. Has any other concurrent anti-cancer therapy (chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational [used for a not approved indication and in the context of a research investigation]) within 28 days of first study drug administration; or plans to participate in an experimental drug study while enrolled in this study.

16. Has any medical contraindications to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Visual and Pathological Response | at 24 weeks
  Visual and pathological response of all treated BCC lesions on participant level assessed by central review

SECONDARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events assessed by CTCAE 5.0 | through study completion, average 7 months
  Occurrence of adverse events (AEs), serious adverse events (SAEs), and AEs leading to discontinuation or death on participant level.
Extent of Pathological Response | at 24 weeks
  Pathological response on participant level assessed by the investigator and central review, respectively, using a 4-point scale
  1. Pathologic Complete Response (pCR): No Residual Viable Tumor (RVT)
  2. Major Pathologic Response (MPR)/ "near-pCR": <= 10% RVT
  3. Pathologic Partial Response (pPR): 10% < RVT <= 50% "
  4. Pathologic Non-Response" (pNR): >50% RVT
Change of Visual Lesion Appearance | at baseline and at 24 weeks
  Visual response [during the study and at surgery] on participant level assessed by the investigator and central review, respectively.
Number of Participants with BCC Recurrence | at 12 and 24 months after surgery
  Recurrence after surgery on participant level assessed by the investigator

CONTACTS AND LOCATIONS:
Locations (10):
- Israel (4):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Hadassah Ein Kerem Medical Center, Jerusalem
  - Kaplan Medical Center, Rehovot
- Spain (6):
  - Hospital Clínic Barcelona, Barcelona
  - Hospital de Basurto, Bilbao
  - Clínica Universitaria de Navarra (CUN), Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Instituto Valenciano de Oncología (IVO), Valencia

IPD SHARING:
Plan to Share IPD: No